CLINICAL TRIAL: NCT04697121
Title: Artichoke and Bergamot Phytosome: a Randomized Double Blind Clinical Trial in Bergamot Poor-responders
Brief Title: Artichoke and Bergamot Phytosome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0921/22052019
Record Dates: First submitted 2020-12-29; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hypercholesterolemia
Keywords: bergamot; Cynara cardunculus
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Combination Product: Placebo
- Combined Bergamot Phytosome and Artichoke leaf dry extract (Active Comparator): 600 mg of Bergamot Phytosome and 100 mg of Artichoke leaf standardized dry extract
  Interventions: Dietary Supplement: Combined Bergamot phytosome and Artichoke leaf dry extract

INTERVENTIONS:
Dietary Supplement: Combined Bergamot phytosome and Artichoke leaf dry extract — 600 mg of Bergamot Phytosome and 100 mg of Artichoke leaf standardized dry extract. Supplementation regimen was 2 daily tablets, one before lunch and one before dinner, for 8 continuous weeks.
  Arms: Combined Bergamot Phytosome and Artichoke leaf dry extract
Combination Product: Placebo — Supplementation regimen was 2 daily tablets, one before lunch and one before dinner, for 8 continuous weeks.
  Arms: Placebo

SUMMARY:
According to WHO data, about 50% of deaths each year are caused by cardiovascular disease. One of the strategies for prevention of cardiovascular diseases, in addition to a correct lifestyle, is to implement therapies that reduce the level of cholesterol in the blood and at the same time control the glycemic levels, which are closely related in the maintenance of metabolic homeostasis. The aim of this clinical study is to confirm the potential broader activity as hypocholesterolemic agent in bergamot poor-responders subjects with mild hypercholesterolemia. The study was a 8-week randomized double-blind placebo-controlled trial. Participants were randomized to either the supplement based on dry extract from artichoke leaf and bergamot phospholipid (31) or placebo arm (29).

ELIGIBILITY:
Inclusion Criteria:

* mild hypercholesterolemia (220 - 280 mg/dl)
* subjects were not taking any medication likely to affect lipid metabolism (such as statins)
* subjects were bergamot poor-responders

Exclusion Criteria:

* liver, renal and thyroid diseases
* history of cardiovascular disease (CVD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Changes of lipid parameters | Baseline / 30 days / 60 days
  Total cholesterol, LDL cholesterol, HDL cholesterol (mg/dl)

SECONDARY OUTCOMES:
Changes of lipid parameters | Baseline / 30 days / 60 days
  apolipoprotein A, apolipoprotein B, triglycerides (mg/dl)
Changes of metabolic parameters | Baseline / 30 days / 60 days
  Fasting blood glucose (mg/dl)
Changes of metabolic parameters | Baseline / 30 days / 60 days
  Glycated Hemoglobin (percent)
Changes of anthropometric measurements | Baseline / 30 days / 60 days
  Weight (kg) and height (m) were combined to report BMI in kg/m^2
Changes of anthropometric measurements | Baseline / 30 days / 60 days
  waist circumference (cm)
Changes of body composition | Baseline / 30 days / 60 days
  Fat mass (g), Fat Free Mass (g), Visceral Adipose Tissue (g)
Changes of safety parameters | Baseline / 30 days / 60 days
  Aspartate Aminotransferase (UI/l), Alanine Aminotransferase (UI/l)
Changes of safety parameters | Baseline / 30 days / 60 days
  Gamma Glutamyl Transferase (U/l)
Changes of safety parameters | Baseline / 30 days / 60 days
  Creatinine (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No